CLINICAL TRIAL: NCT00520429
Title: Transforming Psychotherapy for Chronically Ill Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Cully, Jeffrey - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRECC001
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2008-07

CONDITIONS: Heart Failure, Congestive; Pulmonary Disease, Chronic Obstructive; Depression; Anxiety
Keywords: Depression; Anxiety; Pulmonary Disease, Chronic Obstructive; Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Depression; Anxiety Disorders | interventions — Educational Status; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): This study is an open pilot; therefore all participants were given the opportunity to receive treatment.
  Interventions: Behavioral: ACCES - Adjusting to Chronic Conditions with Education and Support

INTERVENTIONS:
Behavioral: ACCES - Adjusting to Chronic Conditions with Education and Support — The primary objective of this research is to pilot test a brief mental heath treatment specifically tailored to meet the needs of chronically ill patients with anxiety and/or depression. Using an open-trial format, the proposed study will examine the feasibility of a brief psychosocial intervention. Primary outcomes will assess intervention effects on patient and clinician rated symptoms of anxiety and depression. If proven feasible and effective among this group of participants, the intervention (due to its brief format and focus on medically ill patient needs) will possess unique characteristics that will increase the ability of medical care settings to implement mental health treatments, and will provide valuable pilot data for the development of a larger research project to determine the efficacy of this intervention among a larger group of chronically ill patients relative to usual care.

SUMMARY:
The primary objective of this research is to pilot test a brief mental heath treatment specifically tailored to meet the needs of chronically ill patients with anxiety and/or depression. Using an open-trial format, the proposed study will examine the feasibility of a brief psychosocial intervention. Primary outcomes will assess intervention effects on patient and clinician rated symptoms of anxiety and depression. If proven feasible and effective among this group of participants, the intervention (due to its brief format and focus on medically ill patient needs) will possess unique characteristics that will increase the ability of medical care settings to implement mental health treatments, and will provide valuable pilot data for the development of a larger research project to determine the efficacy of this intervention among a larger group of chronically ill patients relative to usual care.

DETAILED DESCRIPTION:
Select one category that most adequately describes your research:

Pilot

Discuss the research design including but not limited to such issues as: probability of group assignment, potential for subject to be randomized to placebo group, use of control subjects, etc.

The proposed project is designed to pilot test the feasibility of a brief psychosocial intervention among depressed and/or anxious medical patients with confirmed symptoms of COPD and/or CHF causing significant impairment as ascertained by validated surveys. We will test the intervention with an open-trial format. Therefore, all patients who meet the inclusion criteria described below will receive the intervention. Group assignment, randomization, and use of control subjects are not applicable to this pilot research project. Data will be collected at baseline, post-treatment (8 weeks), and at 3 month follow-up. Trained members of the study staff will conduct assessments, intervention and follow-up sessions following a protocol. A licensed psychologist will supervise all members of the study staff.

F2. Procedure

Recruitment Procedures: Patients with COPD and CHF who meet criteria for clinically significant physical and emotional symptoms will be recruited. Recruitment of potential participants (detailed further in Section J) will occur through database extractions (e.g. ICD-9 codes), primary care provider referrals, and specialty care provider referrals (e.g. cardiology and pulmonology). Patients will then be contacted via letter, which provides basic information about the study. If no response from the person is received within 5 days, a study research assistant will contact the person via telephone to determine if they are interested and eligible for participation in the study. These procedures are currently being used in related IRB approved studies H#19681 "Mental Health Treatment Engagement In CHF Patients With Depression And Anxiety", and H-19629 "Identifying Mental Health Treatment Barriers in Medically Ill Older Adults".

Telephone Screening: A trained research assistant will administer the 15 minute telephone screen. Prior to the initiation of the telephone screen, patients will be provided with study informed consent and patient verbal assent will be obtained. Following consent, patients will be asked a series of questions to assess: patient information (e.g. demographic data), symptoms of heart failure and/or symptoms of COPD, cognitive functioning (6-item screener), and brief mental health service use history. The RA will also determine eligibility by administering five items from the PRIME-MD to screen for anxiety and depression. Given its high sensitivity to detect depression and anxiety, use of the PRIME-MD will reduce the number of patients without symptoms of depression or anxiety unnecessarily attending in-person interview. If the patient meets study eligibility, they will be invited to attend an in-person study interview.

In-person Screening: Initial screen eligible patients will be invited to an in-person appointment where final eligibility will be determined and baseline assessment measures completed. All appointments will take place at the designated research site. Demographic information will be collected for: age, gender, ethnicity, household income, marital status, education, employment status, and current/past smoking (e.g. pack years). Medical history information will be collected for: date of onset/diagnosis of CHF and/or COPD, current medication usage, and history of other significant illness. The MINI psychiatric interview will be used to determine the presence of DSM-IV Axis I disorders. Symptoms of anxiety and depression will be assessed using self-report and clinician rated instruments to determine final eligibility. Other baseline measures will include assessments for psychiatric diagnoses (semi-structured clinical interview), quality of life (disease specific and general), and health service utilization (by patient self-report). All patients who meet the eligibility requirements described in Section F will be invited to receive the intervention. A study clinician will initiate contact with the patient via telephone and subsequently set up an initial treatment session.

Intervention: The intervention is a psychosocial treatment that was specifically developed to address the mental health and quality of life needs for chronically ill patients. As such the intervention contains a number of unique characteristics that are designed to better address the mental and physical health needs of these patients. It is a skills-based intervention that matches patients' expressed desire for improved quality of life within focused intervention modules based on their symptom profile and preferences for care. Modules are guided by a symptom-based algorithm but ultimately patients choose the intervention focus with the clinician serving as a consultant or guide. All patients receive two core modules focused on increasing awareness and controlling symptoms that emphasizes the overlap and distinction between mental health and physical heath symptoms. At the conclusion of the core modules, patients work with their study clinician to set initial goals for improving quality of life. Goals need not be restricted to "mental health" (e.g. reducing symptoms of depression or anxiety) but can also focus on stress and concerns about their physical condition (e.g. improving functioning and general quality of life by actively coping with a chronic medical illness). Following the core modules, patients are provided with a series of module choices from which they select skills training that matches their current and most pressing needs. Collectively, the active treatment phase is provided over 6 weekly sessions (2 core sessions and 4 elective module sessions). Each session is followed by a brief telephone follow-up that occurs between 1 and 3 days before the next session. At the conclusion of the active treatment phase, the participant will receive three follow-up telephone calls at weeks 8, 10, and 12 (referred to as booster telephone calls) to review skills, encourage continued practice, and facilitate consolidation of treatment gains.

Assessments: Data will be collected at baseline, post-treatment (8 weeks), and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of CHF or COPD diagnosis according to medical chart review
* Ongoing symptoms of functional limitations due to CHF (NYHA classification of II , III, or IV as obtained by telephone interview) or COPD (Score of 3 or greater on the Medical Research Council Dyspnoea Scale [MRC] as obtained by telephone interview)
* Eligible patients must have clinically significant symptoms of either anxiety and/or depression as measured using patient self report questionnaires. Clinical cutoff scores for depression will be based on the Beck Depression Inventory - Second Edition (scores of 14 or more) while anxiety cutoffs will be determined using the State-Trait Anxiety Inventory (score of 40 or greater)
* Eligible patients will be English-speaking, as this intervention has not yet been translated to any other language.

Exclusion Criteria:

* History of substance abuse, bipolar disorder, psychosis or active suicidal intent (obtained from chart review and standardized structured clinical interview)
* NYHA class I, or MRC levels 1 and 2. Class 1 CHF patients and Level 1 and 2 COPD patients (by definition) will have no significantly limiting CHF or COPD symptoms. This information will be obtained through patient self-report of CHF and COPD symptoms
* Mental status examination score in the cognitively impaired range on an established 6-item screen
* Inability to provide informed consent or severe physical limitations restricting completion of the study protocol (e.g. vision, hearing, or physical functioning)
* Non-English speaking patients will be excluded from participation, as this intervention has not yet been translated to any other language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
State-trait Anxiety Inventory (STAI), a 40-item self-report measure of anxiety symptoms.Beck Depression Inventory-II (BDI-II), assessing 21 depression symptoms. Client Satisfaction Questionnaire (CSQ), an 8-item, empirical, self-report measure. | Assessments at baseline, post treatment, and 3 month follow-up.

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ), a 23-item self-report measure of constructs. Chronic Respiratory Questionnaire (CRQ), measuring QoL change over time in COPD patients. Short Form 36 (SF-36), a generic measure of health-related QoL. | Assessments at baseline, post treatment, and 3 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cully, PhD MEd BS, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Houston VA Medical Center, Houston, Texas, United States